CLINICAL TRIAL: NCT05712603
Title: A Care Path for the Detection of Advanced NAFLD-fibrosis: the Nijmegen-Leiden-Amsterdam 2-tiered Care Path Study - the NLA2 Study
Brief Title: The Nijmegen-Leiden-Amsterdam 2-tiered Care Path Study
Acronym: NLA2
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Maag Lever Darm Stichting (Other); Radboud University Medical Center (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Onno Holleboom, MD, PhD, Vascular internist and endocrinologist, Assistant professor, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL81357.018.22
Record Dates: First submitted 2022-10-19; First posted 2023-02-03 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Care path; Non-alcoholic Fatty Liver Disease; FIB4; FibroScan; ELF-test
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum of the participants will be retained if they give permission for that. buffy coats will be stored as well, for future DNA research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prospective care path arm: Participants who enter the care path will make up the prospective care path arm.
  In patients entering the care path three diagnostic tests for liver fibrosis will be performed. FIB4-score, Vibration controlled transient elastography and Enhanced Liver Fibrosis test
  Interventions: Diagnostic Test: FIB4-score; Diagnostic Test: Vibration controlled transient elastography; Diagnostic Test: Enhanced Liver Fibrosis test
- Prospective arm of 'regular care': Patients who are referred to the hepatologist in participating centers during the study period without using the care path (e.g. because of altered liver function tests for instance), will be the prospective 'regular care' arm
- Retrospective arm of 'regular care': The investigators will do an data extraction of the electronic health records of patients referred to the hepatologist in the five years prior to the study. They will make up the retrospective comparative arm of regular care

INTERVENTIONS:
Diagnostic Test: FIB4-score — A score which estimates the risk for advanced liver fibrosis, based on: age, ALT, AST and thrombocytes
  Groups: Prospective care path arm
Diagnostic Test: Vibration controlled transient elastography — VCTE measures the speed of a mechanically generated shear wave across the liver to derive a liver stiffness measurement (LSM), a marker of hepatic fibrosis
  Other Names: VCTE
  Groups: Prospective care path arm
Diagnostic Test: Enhanced Liver Fibrosis test — The ELF-test is a non-invasive blood test that measures three direct markers of liver fibrosis: hyaluronic acid (HA), procollagen III amino-terminal peptide (PIIINP), and tissue inhibitor of matrix metalloproteinase 1 (TIMP-1).
  Other Names: ELF-test
  Groups: Prospective care path arm

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a liver disease, caused by storage of fat in the liver. The most-important risk-factors are being overweight, and disorders in sugar and cholesterol handling of the body. On average does around 30% of the population worldwide have any signs of fatty liver. Most people will not get severe complaints as a result of their fatty liver. But in some of them, the fat storage will lead to hepatitis. This causes damage to the liver which can eventually lead to scarring of the liver, and in some patients to cirrhosis. This possibly can cause liver failure, liver cancer, an several complaints which reduce the quality of life. There are several tests which can help in detecting scarring of the liver. However, the scientific world still does not know well enough which test works best and if they perhaps might work better if they are used together. In this study these questions will be investigated in order to design a care path which does several tests consecutively. The goal is that this will make it possible to easily detect a severely diseased liver and that this will eventually help to detect patients earlier so they can be treated earlier and complications of the disease might be reduced. Moreover, is the goal that this study will lead to a decrease in unnecessary referrals to a hepatologist, resulting in a reduction in invasive diagnostic interventions. Hospital specialists who think that their patient might be at risk for advanced liver disease, can refer a patient to this study. Participants will go to the hospital for one study visit where several tests will be done which are designed to detect liver scarring. Depending on the results, a participant will be referred to a hepatologist for more extensive diagnostics or referred back to the referring specialist with advice for management of the disease.

DETAILED DESCRIPTION:
Background of the study:

Non-alcoholic fatty liver disease (NAFLD) is a disease of alarmingly increasing prevalence. Progression along the NAFLD spectrum often goes unnoticed since it is often asymptomatic. Awareness among health care workers and implementation of care paths to detect progressing NAFLD stages are limited. Without clear guidance papers or robust care pathways for risk stratification, the current diagnostic approach for NAFLD is highly variable, leading to both underdiagnosis of advanced stages of disease, andunnecessary referrals for mild stages of disease. This calls for a comprehensive care path consisting of non-invasive alternatives to detect those patients with severe cases of NAFLD. Particularly the use of a sequential, two-tiered care path algorithm is promising as it has the ability to detect underlying advanced cases of fibrosis, and has previously been shown to be cost-effective. This was shown by dr. Ankur Srivastava, who designed a pathway consisting of FIB4-score and ELF-test that led to a reduction of unnecessary referrals to the hepatologist by 80%, whilst improving the detection of advanced fibrosis and cirrhosis 5- and 3-fold,respectively (8). In this study the investigation of several two-tiered sequential care path algorithms, comprised of the FIB4-score, VCTE and the ELF-test, for the detection of advanced stages of NAFLD-fibrosis is proposed: the Nijmegen-Leiden-AmsterdamNAFLD-NASH 2-tiered care path study: NLA2-study.

Objective of the study:

The aim of the study is to improve case finding of advanced cases of NAFLD (≥F3 fibrosis), whilst simultaneously reducing unnecessary referrals for mild cases (<F3 fibrosis). Additionally, the aim is to increase awareness of NAFLD, and NAFLD-related complications, and to assess the cost-effectiveness of the different proposed care paths compared to current regular care.

Study design:

This is a care innovation study, with an estimated duration of three years. The intend is to commence the study at three academic medical centres namely in Nijmegen, Leiden and Amsterdam, with the intention to include other non-academic hospitals after the initial roll-out. The study has both a prospective and a retrospective part. The prospective part consists of participants who are deemed by their treating specialist physician to be at risk of severe NASH fibrosis. Participants will be invited to attend a study visit.

This study visit will consist of, among others: anthropometric measurements, blood pressure measurement, blood sampling and VCTE. The diagnostic testing for potentially underlying advanced (≥F3) liver fibrosis consists of the FIB4-score, VCTE and the ELF-test. A blood sample will be stored for additional biomarker testing. Based on predefined cut-offs for the FIB4-score and liver stiffness measurement (LSM) (measured using VCTE), participants will be classified as being at low or high risk of advanced (≥F3)fibrosis (see figure 1). The ELF-test will be analysed in bulk and will thus not be used for risk assessment. Participants classified at low risk will remain under the care of their treating specialist. Participants classified at high risk of advanced (≥F3) fibrosis will be referred to a hepatologist. Read-outs of the electronic health records (EHR) of all participants will be performed at 24 months after inclusion in the study, an dat six months for those classified at high risk. Read-outs will be performed to assess the correctness of the risk assessment and subsequent referral to the hepatologist.

The three different sequential, two-tiered care path algorithms will be evaluated upon completion of the study. The diagnostic accuracy, defined as sensitivity, specificity, predictive values and AUROCs, of the three different care path algorithms will be calculated. The diagnostic performance will be expressed as the percentage of correct referrals and the percentage of unnecessary referrals of the different care path algorithms and the individual non-invasive tests, compared to regular care.

Study population:

The study population consists of adults (≥ 18 years old) who are suspected by their treating specialist to suffer from a severe stage of NAFLD-fibrosis. Exclusion criteria are, most notably, a previous diagnosis of advanced (≥F3) fibrosis, any other known chronic liver disease, use of drugs that may cause drug-induced steatosis, and present excessive alcohol use. The aim is to include 200 patients in analyses in total, of which 100 will be referred using the NLA2 study and 100 through regular care. The latter group will form the prospective comparator arm. This necessitates a 50% adherence rate of participating hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Suspected by treating physician to suffer from a severe stage of NAFLD-fibrosis.

Exclusion Criteria:

* Previous diagnosis of advanced (≥F3) liver fibrosis;
* Any other known chronic liver disease (alcoholic steatohepatitis, hepatitis B, hepatitis C, autoimmune hepatitis, hemochromatosis, Wilsons disease, alpha-1-antitrypsin deficiency);
* Drugs that may cause drug-induced hepatic steatosis, (table provided elsewhere)
* Present excessive alcohol use, defined as > 2 units/day for women and > 3 units/day for men;
* A psychiatric, addictive or any other disorder that compromises the subject's ability to understand the study content and to give written informed consent for the participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from three different academic medical centres in the Netherlands, namely Radboudumc, LUMC and Amsterdam UMC. Patients who are suspected of underlying severe NAFLD-fibrosis by their treating physician are eligible for inclusion in the study. This suspection will most often arise because of risk factors as obesity, diabetes type 2, hypercholesterolemia or metabolic syndrome, or proven heaptic steatosis because of an conventional ultrasound. Patients are referred from hospital specialists
Sampling Method: Non-Probability Sample
Enrollment: 655 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the three different care paths to detect advanced fibrosis. | The time frame is based on the time between the study visit and the subsequent read-outs of the EHR, up to 24 months later
  The diagnostic accuracy of the three different sequential care path algorithms to detect underlying advanced (≥F3) liver fibrosis, assessed using sensitivity, specificity, predictive values and area under the receiver characteristics (AUROC) curve
Diagnostic performance of the three different care paths to increase correct and decrease incorrect referrals. | The time frame is based on the time between the study visit and the subsequent read-outs of the EHR, up to 24 months later
  The diagnostic performance of the three different sequential care path algorithms, defined as the increase in correct and the decrease in unnecessary referrals when using these care paths to detect underlying advanced (≥F3) NAFLD-fibrosis compared to regular care.

SECONDARY OUTCOMES:
Cost effectiveness of the different diagnostic modalities/care path algorithms | The time frame is based on the time between the study visit and the subsequent read-outs of the EHR, up to 24 months later.
  The cost effectiveness of the different diagnostic modalities/care path algorithms compared to each other and to regular care.
Number of patients coded for NAFLD before and after the study | through study completion, an average of 1 year
  Number of patients coded for NAFLD by physicians before and after initiation of the NLA2 study (measure of awareness)
The diagnostic accuracy of the FIB4-score for detecting advanced fibrosis | The time frame is based on the time between the study visit and the subsequent read-outs of the EHR, up to 24 months later.
  The diagnostic accuracy of the FIB4-score for detecting underlying advanced (≥F3) liver fibrosis, using sensitivity, specificity, predictive values and AUROC-curves;
The diagnostic accuracy of the ELF-test for detecting advanced fibrosis | The time frame is based on the time between the study visit and the subsequent read-outs of the EHR, up to 24 months later.
  The diagnostic accuracy of the ELF-test for detecting underlying advanced (≥F3) liver fibrosis, using sensitivity, specificity, predictive values and AUROC-curves;
The diagnostic accuracy of VCTE for detecting advanced fibrosis | The time frame is based on the time between the study visit and the subsequent read-outs of the EHR, up to 24 months later.
  The diagnostic accuracy of VCTE for detecting underlying advanced (≥F3) liver fibrosis, using sensitivity, specificity, predictive values and AUROC-curves;
Diagnostic performance of the FIB4-score to increase correct and decrease incorrect referrals. | The time frame is based on the time between the study visit and the subsequent read-outs of the EHR, up to 24 months later.
  The diagnostic performance of the FIB4-score, defined as the increase in correct and the decrease in unnecessary referrals when using this test to detect underlying advanced (≥F3) NAFLD-fibrosis compared to regular care.
Diagnostic performance of VCTE to increase correct and decrease incorrect referrals. | The time frame is based on the time between the study visit and the subsequent read-outs of the EHR, up to 24 months later.
  The diagnostic performance of VCTE, defined as the increase in correct and the decrease in unnecessary referrals when using this test to detect underlying advanced (≥F3) NAFLD-fibrosis compared to regular care.
Diagnostic performance of the ELF-test to increase correct and decrease incorrect referrals. | The time frame is based on the time between the study visit and the subsequent read-outs of the EHR, up to 24 months later.
  The diagnostic performance of the ELF-test, defined as the increase in correct and the decrease in unnecessary referrals when using this test to detect underlying advanced (≥F3) NAFLD-fibrosis compared to regular care.

CONTACTS AND LOCATIONS:
Overall Officials: Onno Holleboom, MD PhD, Principal Investigator — Amsterdam UMC, location AMC
Locations (3):
- Netherlands (3):
  - Radboudumc, Nijmegen, Gelderland
  - Amsterdam UMC, location AMC, Amsterdam, North Holland
  - Leiden universitair medisch centrum, Leiden, South Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stols-Goncalves D, Hovingh GK, Nieuwdorp M, Holleboom AG. NAFLD and Atherosclerosis: Two Sides of the Same Dysmetabolic Coin? Trends Endocrinol Metab. 2019 Dec;30(12):891-902. doi: 10.1016/j.tem.2019.08.008. Epub 2019 Oct 17. PMID 31630897
- [Background] Tushuizen ME, Holleboom AG, Koot BGP, Blokzijl H, van Mil SWC, Koek GH. [Non-alcoholic fatty liver disease; a full-bodied epidemic]. Ned Tijdschr Geneeskd. 2020 Feb 27;164:D4096. Dutch. PMID 32267638
- [Background] Lazarus JV, Ekstedt M, Marchesini G, Mullen J, Novak K, Pericas JM, Roel E, Romero-Gomez M, Ratziu V, Tacke F, Cortez-Pinto H, Anstee QM; EASL International Liver Foundation NAFLD Policy Review Collaborators. A cross-sectional study of the public health response to non-alcoholic fatty liver disease in Europe. J Hepatol. 2020 Jan;72(1):14-24. doi: 10.1016/j.jhep.2019.08.027. Epub 2019 Sep 10. PMID 31518646
- [Background] Harris R, Harman DJ, Card TR, Aithal GP, Guha IN. Prevalence of clinically significant liver disease within the general population, as defined by non-invasive markers of liver fibrosis: a systematic review. Lancet Gastroenterol Hepatol. 2017 Apr;2(4):288-297. doi: 10.1016/S2468-1253(16)30205-9. Epub 2017 Feb 1. PMID 28404158
- [Background] Crossan C, Tsochatzis EA, Longworth L, Gurusamy K, Davidson B, Rodriguez-Peralvarez M, Mantzoukis K, O'Brien J, Thalassinos E, Papastergiou V, Burroughs A. Cost-effectiveness of non-invasive methods for assessment and monitoring of liver fibrosis and cirrhosis in patients with chronic liver disease: systematic review and economic evaluation. Health Technol Assess. 2015 Jan;19(9):1-409, v-vi. doi: 10.3310/hta19090. PMID 25633908
- [Background] Tapper EB, Sengupta N, Hunink MG, Afdhal NH, Lai M. Cost-Effective Evaluation of Nonalcoholic Fatty Liver Disease With NAFLD Fibrosis Score and Vibration Controlled Transient Elastography. Am J Gastroenterol. 2015 Sep;110(9):1298-304. doi: 10.1038/ajg.2015.241. Epub 2015 Aug 25. PMID 26303130
- [Background] Srivastava A, Gailer R, Tanwar S, Trembling P, Parkes J, Rodger A, Suri D, Thorburn D, Sennett K, Morgan S, Tsochatzis EA, Rosenberg W. Prospective evaluation of a primary care referral pathway for patients with non-alcoholic fatty liver disease. J Hepatol. 2019 Aug;71(2):371-378. doi: 10.1016/j.jhep.2019.03.033. Epub 2019 Apr 6. PMID 30965069
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Estes C, Razavi H, Loomba R, Younossi Z, Sanyal AJ. Modeling the epidemic of nonalcoholic fatty liver disease demonstrates an exponential increase in burden of disease. Hepatology. 2018 Jan;67(1):123-133. doi: 10.1002/hep.29466. Epub 2017 Dec 1. PMID 28802062
- [Background] Younossi Z, Anstee QM, Marietti M, Hardy T, Henry L, Eslam M, George J, Bugianesi E. Global burden of NAFLD and NASH: trends, predictions, risk factors and prevention. Nat Rev Gastroenterol Hepatol. 2018 Jan;15(1):11-20. doi: 10.1038/nrgastro.2017.109. Epub 2017 Sep 20. PMID 28930295
- [Background] Ruissen MM, Mak AL, Beuers U, Tushuizen ME, Holleboom AG. Non-alcoholic fatty liver disease: a multidisciplinary approach towards a cardiometabolic liver disease. Eur J Endocrinol. 2020 Sep;183(3):R57-R73. doi: 10.1530/EJE-20-0065. PMID 32508312
- [Background] Taylor RS, Taylor RJ, Bayliss S, Hagstrom H, Nasr P, Schattenberg JM, Ishigami M, Toyoda H, Wai-Sun Wong V, Peleg N, Shlomai A, Sebastiani G, Seko Y, Bhala N, Younossi ZM, Anstee QM, McPherson S, Newsome PN. Association Between Fibrosis Stage and Outcomes of Patients With Nonalcoholic Fatty Liver Disease: A Systematic Review and Meta-Analysis. Gastroenterology. 2020 May;158(6):1611-1625.e12. doi: 10.1053/j.gastro.2020.01.043. Epub 2020 Feb 4. PMID 32027911
- [Background] Dulai PS, Singh S, Patel J, Soni M, Prokop LJ, Younossi Z, Sebastiani G, Ekstedt M, Hagstrom H, Nasr P, Stal P, Wong VW, Kechagias S, Hultcrantz R, Loomba R. Increased risk of mortality by fibrosis stage in nonalcoholic fatty liver disease: Systematic review and meta-analysis. Hepatology. 2017 May;65(5):1557-1565. doi: 10.1002/hep.29085. Epub 2017 Mar 31. PMID 28130788
- [Background] Sumida Y, Nakajima A, Itoh Y. Limitations of liver biopsy and non-invasive diagnostic tests for the diagnosis of nonalcoholic fatty liver disease/nonalcoholic steatohepatitis. World J Gastroenterol. 2014 Jan 14;20(2):475-85. doi: 10.3748/wjg.v20.i2.475. PMID 24574716
- [Background] Alexander M, Loomis AK, van der Lei J, Duarte-Salles T, Prieto-Alhambra D, Ansell D, Pasqua A, Lapi F, Rijnbeek P, Mosseveld M, Avillach P, Egger P, Dhalwani NN, Kendrick S, Celis-Morales C, Waterworth DM, Alazawi W, Sattar N. Non-alcoholic fatty liver disease and risk of incident acute myocardial infarction and stroke: findings from matched cohort study of 18 million European adults. BMJ. 2019 Oct 8;367:l5367. doi: 10.1136/bmj.l5367. PMID 31594780
- [Background] Graupera I, Thiele M, Serra-Burriel M, Caballeria L, Roulot D, Wong GL, Fabrellas N, Guha IN, Arslanow A, Exposito C, Hernandez R, Aithal GP, Galle PR, Pera G, Wong VW, Lammert F, Gines P, Castera L, Krag A; Investigators of the LiverScreen Consortium. Low Accuracy of FIB-4 and NAFLD Fibrosis Scores for Screening for Liver Fibrosis in the Population. Clin Gastroenterol Hepatol. 2022 Nov;20(11):2567-2576.e6. doi: 10.1016/j.cgh.2021.12.034. Epub 2021 Dec 29. PMID 34971806
- [Background] Marjot T, Moolla A, Cobbold JF, Hodson L, Tomlinson JW. Nonalcoholic Fatty Liver Disease in Adults: Current Concepts in Etiology, Outcomes, and Management. Endocr Rev. 2020 Jan 1;41(1):bnz009. doi: 10.1210/endrev/bnz009. PMID 31629366
- [Background] Eddowes PJ, Sasso M, Allison M, Tsochatzis E, Anstee QM, Sheridan D, Guha IN, Cobbold JF, Deeks JJ, Paradis V, Bedossa P, Newsome PN. Accuracy of FibroScan Controlled Attenuation Parameter and Liver Stiffness Measurement in Assessing Steatosis and Fibrosis in Patients With Nonalcoholic Fatty Liver Disease. Gastroenterology. 2019 May;156(6):1717-1730. doi: 10.1053/j.gastro.2019.01.042. Epub 2019 Jan 25. PMID 30689971
- [Background] Siddiqui MS, Vuppalanchi R, Van Natta ML, Hallinan E, Kowdley KV, Abdelmalek M, Neuschwander-Tetri BA, Loomba R, Dasarathy S, Brandman D, Doo E, Tonascia JA, Kleiner DE, Chalasani N, Sanyal AJ; NASH Clinical Research Network. Vibration-Controlled Transient Elastography to Assess Fibrosis and Steatosis in Patients With Nonalcoholic Fatty Liver Disease. Clin Gastroenterol Hepatol. 2019 Jan;17(1):156-163.e2. doi: 10.1016/j.cgh.2018.04.043. Epub 2018 Apr 26. PMID 29705261
- [Background] Vali Y, Lee J, Boursier J, Spijker R, Loffler J, Verheij J, Brosnan MJ, Bocskei Z, Anstee QM, Bossuyt PM, Zafarmand MH; LITMUS systematic review team(dagger). Enhanced liver fibrosis test for the non-invasive diagnosis of fibrosis in patients with NAFLD: A systematic review and meta-analysis. J Hepatol. 2020 Aug;73(2):252-262. doi: 10.1016/j.jhep.2020.03.036. Epub 2020 Apr 8. PMID 32275982
- [Background] Younossi ZM, Golabi P, de Avila L, Paik JM, Srishord M, Fukui N, Qiu Y, Burns L, Afendy A, Nader F. The global epidemiology of NAFLD and NASH in patients with type 2 diabetes: A systematic review and meta-analysis. J Hepatol. 2019 Oct;71(4):793-801. doi: 10.1016/j.jhep.2019.06.021. Epub 2019 Jul 4. PMID 31279902
- [Background] Nabi O, Lacombe K, Boursier J, Mathurin P, Zins M, Serfaty L. Prevalence and Risk Factors of Nonalcoholic Fatty Liver Disease and Advanced Fibrosis in General Population: the French Nationwide NASH-CO Study. Gastroenterology. 2020 Aug;159(2):791-793.e2. doi: 10.1053/j.gastro.2020.04.048. Epub 2020 May 4. No abstract available. PMID 32376412